CLINICAL TRIAL: NCT01834404
Title: Peripheral Pharmacodynamics of Phentermine-Topiramate in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, Primary Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-000948; R01DK067071 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2013-03-27; First posted 2013-04-17 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
Keywords: Obesity; BMI; Incretin; Satiety; Phentermine; Topiramate
MeSH Terms: conditions — Obesity | interventions — Qsymia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phentermine-Topiramate ER (Experimental): Qualifying participants were assigned to the Phentermine-Topiramate ER for a minimum of 5 days. The dosing of the study drug was phentermine 3.75 mg / topiramate 23 mg days 1-5. The dosing of the study drug was increased to phentermine 7.5 mg / topiramate 46 mg days 6-14.
  Interventions: Drug: Phentermine-Topiramate ER
- Placebo (Placebo Comparator): Qualifying participants were assigned to placebo for a minimum of 5 days. Placebo pills matched the study drug in appearance for the 2 dose levels.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phentermine-Topiramate ER — The dosing of the study drug was phentermine 3.75 mg / topiramate 23 mg days 1-5. The dosing of the study drug was increased to phentermine 7.5 mg / topiramate 46 mg days 6-14.
  Other Names: Qsymia
  Arms: Phentermine-Topiramate ER
Drug: Placebo — Placebo pills matched the study drug in appearance for the 2 dose levels.
  Arms: Placebo

SUMMARY:
Our overall goal is to determine the effect of Phentermine and Topiramate ER on gastric emptying, gastric accommodation, satiety, and satiation in obese participants.

DETAILED DESCRIPTION:
Investigators propose a randomized controlled trial of combination phentermine topiramate ER versus placebo given orally for 10-15 days.

At visit 1 subjects had a brief interview, body measurements, and completed 4 questionnaires to rule out any gastrointestinal or significant psychological distress.

At visit 2 subjects did a satiation/nutrient drink test. They drank a nutrient drink until they reached the maximum volume that could be tolerated, symptoms were recorded and blood samples taken at 4 times. They were randomized to one of the arms, and received a 5 day supply of study medication or placebo. The dosing of the study drug was phentermine 3.75 mg / topiramate 23 mg days 1-5.

At visit 3 subjects returned to pick up a nine day supply of study medication or placebo. The dosing of the study drug was increased to phentermine 7.5 mg / topiramate 46 mg days 6-14.

At visit 4 subjects underwent imaging to measure the volume of their stomach with an external camera that revolved around abdomen while they were lying on a table. Stomach volume was checked during fasting, starting 10 min after an intravenous injection of a radioactive material. The subjects ingested more of the liquid nutrient drink and 2 more images were obtained over 30 minutes. On the same day, subjects participated in an all you can eat meal, starting 4 hours after the ingestion of the liquid nutrient drink.

At visit 5 subjects repeated the satiation/nutrient drink test. They drank a nutrient drink until they reached the maximum volume that could be tolerated, symptoms were recorded and blood samples taken at 4 times.

At visit 6 subjects took part in a gastric emptying by scintigraphy test. Subjects were given a scrambled egg breakfast with toast and a glass of milk. The eggs and milk contained a small amount of radioactive substance. At the completion of the meal, subjects stood in front of a special camera and pictures were taken at specific intervals.

ELIGIBILITY:
INCLUSION CRITERIA:

* Obese subjects with BMI> 30 Kg/m^2. Otherwise healthy individuals who are not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrine (other than hyperglycemia not requiring medical therapy) and unstable psychiatric disease.
* Women of childbearing potential will have negative pregnancy test before initiation of medication.

EXCLUSION CRITERIA:

* Weight >300 lbs, which is the limit of safety for the SPECT scanner
* Concomitant use of appetite suppressants (i.e., caffeine based or diethylpropion) or orlistat (Xenical®)
* Uncontrolled hypertension (Blood pressure greater than 160/90 mmHg)
* Concentration of fasting glucose greater than 240 mg/dl
* Concentration of triglycerides greater than 400 mg/dl
* Type 1 Diabetes
* Use of anti-diabetic drugs other than metformin,
* History of nephrolithiasis,
* Recurrent major depression, presence or history of suicidal behavior or ideation with intent to act, and current substantial depressive symptoms (Patient Health Questionnaire-9, 21 total score ≥10).
* Concomitant use of Monoamine Oxidase Inhibitors (MAOI) (i.e., phenelzine, selegiline), serotonergic agents, and other centrally acting appetite suppressants
* Significant psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Scale [HADS] self-administered alcoholism screening test (SAAST, substance abuse) and the questionnaire on eating and weight patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a Hospital Anxiety and Depression Scale (HADS) score ≥11 in any of the subscales or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* End stage renal disease or liver cirrhosis
* Intake of medication that could interfere with the interpretation of the study or cause drug interaction (i.e., ketoconazole, erythromycin). Specifically, birth control pill, estrogen replacement therapy, and thyroxine replacement are permissible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Acosta A, Camilleri M, Shin A, Vazquez-Roque MI, Iturrino J, Burton D, O'Neill J, Eckert D, Zinsmeister AR. Quantitative gastrointestinal and psychological traits associated with obesity and response to weight-loss therapy. Gastroenterology. 2015 Mar;148(3):537-546.e4. doi: 10.1053/j.gastro.2014.11.020. Epub 2014 Dec 6. PMID 25486131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients attending the Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Phentermine-Topiramate ER | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phentermine-Topiramate ER | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (1.8) | 38.2 (2.4) | 34.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat. A body mass index of under 20 is considered to be underweight, while a body mass index between 20 to 25 is considered healthy. A body mass index in the range of 25 to 30 is regarded as overweight. A body mass index over 30 is regarded as obese.
  kg/m^2 | 35.8 (0.9) | 33.9 (1.9) | 34.9 (5.1)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 108.5 (2.2) | 111.2 (2.2) | 109.8 (7.5)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 94.2 (2.7) | 96.5 (3.6) | 95.3 (10.6)
Baseline Volume to Fullness [Mean (Standard Deviation); unit: ml] — At visit 2, subjects did a satiation/nutrient drink test. Participants recorded their sensations every 5 minutes using a numerical scale from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This baseline measure is the volume consumed when the fullness sensation reached level 3.
  ml | 712 (86) | 710 (95) | 711.3 (306.3)
Baseline Maximum Tolerated Volume [Mean (Standard Deviation); unit: ml] — At visit 2, subjects did a satiation/nutrient drink test. Participants recorded their sensations every 5 minutes using a numerical scale from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This baseline measure is the volume consumed when the fullness sensation reached level 5.
  ml | 1368 (111) | 1227 (111) | 1297.8 (383.2)

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying of Solids Half-Time (T 1/2)
Description: Gastric emptying of solids half-time is defined as the time for half of the ingested solids to leave the stomach. At visit 6 subjects took part in a gastric emptying by scintigraphy test. Subjects were given a scrambled egg breakfast with toast and a glass of milk. The eggs and milk contained a small amount of radioactive substance. At the completion of the meal, subjects stood in front of a special camera and pictures were taken at specific intervals.
Time Frame: Day 15, approximately 2 hours after radiolabeled meal was ingested
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
minutes | 109 (7) | 88 (7)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.057, ANCOVA

2. Secondary Outcome: Solid Gastric Emptying: Proportion of Meal Emptied at 2 Hours
Description: At visit 6 subjects took part in a gastric emptying by scintigraphy test. Subjects were given a scrambled egg breakfast with toast and a glass of milk. The eggs and milk contained a small amount of radioactive substance. At the completion of the meal, subjects stood in front of a special camera and pictures were taken at specific intervals. This outcome measure is the proportion of the radiolabeled meal emptied at 2 hours.
Time Frame: Day 15, approximately 2 hours after radiolabeled meal was ingested
Measure: Least Squares Mean (Standard Error); unit: proportion of meal emptied
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
proportion of meal emptied | 0.56 (0.03) | 0.66 (0.03)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.052, ANCOVA

3. Primary Outcome: Fasting Gastric Volume
Description: Fasting whole gastric volume was measured by Technetium (99mTc)-SPECT Imaging. Subjects reported to the clinic after an overnight fast. 99mTC was given by an intravenous injection in the forearm. Tomographic images of the gastric wall were obtained throughout the long axis of the stomach using a dual-head gamma camera that rotates around the body. This allows assessment of the radiolabeled circumference of the gastric wall, rather than the intragastric content.
Time Frame: Day 13, approximately 10 minutes after Technetium (99mTC) injection
Measure: Mean (Standard Error); unit: mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
mL | 227 (25) | 261 (25)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.36, ANCOVA

4. Primary Outcome: Postprandial Gastric Volume
Description: Postprandial gastric volume was measured by 99mTc-SPECT Imaging. Subjects reported to the clinic after an overnight fast. 99mTC was given by an intravenous injection in the forearm. After the liquid meal tomographic images of the gastric wall were obtained throughout the long axis of the stomach using a dual-head gamma camera that rotates around the body. This allows assessment of the radiolabeled circumference of the gastric wall, rather than the intragastric content.
Time Frame: Day 13, approximately 30 minutes after liquid meal
Measure: Mean (Standard Error); unit: mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
mL | 680 (37) | 681 (37)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.99, ANCOVA

5. Primary Outcome: Volume to Fullness
Description: At visit 5, subjects did a satiation/nutrient drink test. Participants recorded their sensations every 5 minutes using a numerical scale from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This measure was the volume consumed when the fullness sensation reached level 3.
Time Frame: Day 14, approximately 30 minutes after liquid meal
Measure: Mean (Standard Error); unit: mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
mL | 570 (63.2) | 630 (61.1)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.45, ANCOVA

6. Primary Outcome: Maximum Tolerated Volume
Description: At visit 5, subjects did a satiation/nutrient drink test. Participants recorded their sensations every 5 minutes using a numerical scale from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This measure is the volume consumed when the fullness sensation reached level 5.
Time Frame: Day 14, approximately 30 minutes after liquid meal
Measure: Mean (Standard Error); unit: mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
mL | 966 (79) | 1108 (79)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.22, ANCOVA

7. Primary Outcome: Buffet Meal Intake
Description: At visit 4 subjects underwent imaging to measure the volume of their stomach, fasting and after ingesting a liquid nutrient drink. Four hours after the liquid meal, subjects were invited to eat, over a 30-minute period, a standard "all you can eat" meal vegetable lasagna, vanilla pudding, and skim milk. The total Kcal of the food consumed was analyzed by using validated software.
Time Frame: Day 13, approximately 4.5 hours after liquid meal
Measure: Mean (Standard Error); unit: Kcal
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
Kcal | 728 (79) | 988 (79)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.032, ANCOVA

8. Secondary Outcome: Solid Gastric Emptying: Proportion Remaining at 4 Hours
Description: At visit 6 subjects took part in a gastric emptying by scintigraphy test. Subjects were given a scrambled egg breakfast with toast and a glass of milk. The eggs and milk contained a small amount of radioactive substance. At the completion of the meal, subjects stood in front of a special camera and pictures were taken at specific intervals. This outcome measure is the proportion of the radiolabeled meal remaining at 4 hours.
Time Frame: Day 15, approximately 4 hours after radiolabeled meal was ingested
Measure: Least Squares Mean (Standard Error); unit: proportion of meal remaining
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
proportion of meal remaining | 0.09 (0.02) | 0.16 (0.02)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; This p-value was based on a rank transformation; Test type: Superiority or Other; p = 0.030, ANCOVA

9. Secondary Outcome: Change in Postprandial Gastric Volume
Description: Change between postprandial and fasting whole gastric volume by 99mTc-SPECT Imaging. A noninvasive SPECT method was used to measure gastric volume during fasting and 32 min after a liquid nutritional supplement meal. Subjects reported to the clinic after an overnight fast. 99mTC was given by an intravenous injection in the forearm. The first fasting scan was obtained, and the study medication was given s.c. After 10 min, a 2nd fasting post medication scan was obtained, and the meal consumed; then two serial postprandial scans were obtained. Each scan required 9-12 min. Tomographic images of the gastric wall were obtained throughout the long axis of the stomach using a dual-head gamma camera that rotates around the body. This allows assessment of the radiolabeled circumference of the gastric wall, rather than the intragastric content.
Time Frame: Day 13, approximately approximately 30 min after liquid meal
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
mL | 453 (24) | 420 (24)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.35, ANCOVA

10. Secondary Outcome: Fasting Ghrelin
Description: Plasma gastrointestinal hormone total ghrelin was measured by radioimmunoassay.
Time Frame: Day 14, before liquid meal
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL | 78.1 (5.6) | 82.6 (10.8)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.72, ANCOVA

11. Secondary Outcome: Peak Postprandial Level of Cholecystokinin (CCK)
Description: Plasma gastrointestinal hormone CCK was measured by radioimmunoassay based on an antibody with very low cross-reactivity to gastrin 17 and its sulfated counterpart, and to sensitivity to a concentration of 0.3 pmol/L.
Time Frame: Day 14, approximately 45 minutes after liquid meal
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL | 8.1 (0.9) | 8.3 (1)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.90, ANCOVA

12. Secondary Outcome: Peak Postprandial Level of Total Glucagon-Like Peptide-1 (GLP-1)
Description: Plasma gastrointestinal hormone GLP-1 was measured by radioimmunoassay.
Time Frame: Day 14, approximately 45 minutes after liquid meal
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL | 13.0 (1.8) | 11.9 (1.6)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.54, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Peak Postprandial Level of Total Peptide Tyrosine-Tyrosine (PYY)
Description: Plasma gastrointestinal hormone PYY was measured by radioimmunoassay.
Time Frame: Day 14, approximately 45 minutes after liquid meal
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Phentermine-Topiramate ER | Placebo
Number analyzed (Participants) | 12 | 12
pg/mL | 195.3 (21.2) | 166 (15.7)
Statistical Analysis 1: Comparison: Phentermine-Topiramate ER vs Placebo; Test type: Superiority or Other; p = 0.26, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Phentermine-Topiramate ER | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes